CLINICAL TRIAL: NCT06706778
Title: Impacts of Music-based Intervention on Pain in Individuals With Irritable Bowel Syndrome (IBS): A Mechanistic Pilot Study
Brief Title: The Mechanism Underlying the Analgesic Effect of the Music of IBS Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000039033
Record Dates: First submitted 2024-11-20; First posted 2024-11-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Abdominal Pain/ Discomfort; Irritable Bowel Syndrome
Keywords: abdominal pain; Music; Brain-gut axis; Stress; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Intervention Model Description: Based on the NIH toolkit and MBIs reporting guidelines, the engagement in this pilot study will be receptive by providing participants with prerecorded, preselected playlists. Participants will also receive a guided video on maximizing music's therapeutic benefits. The playlists will be purely instrumental, with a 60-80 bpm tempo, and feature melodies and harmonies designed for stress relief, including soothing, grounding, meditation, emotional release, etc. This approach is resource-efficient and easily accessible, allowing participants to integrate it into daily pain self-management strategies. Participants will be asked to engage in the MBI in the morning and at night for 30 minutes each, wearing the abdominal belt and smartwatch.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music group (Experimental): Based on the NIH toolkit and MBIs reporting guidelines, the engagement in this pilot study will be receptive by providing participants with prerecorded, preselected playlists. Participants will also receive a guided video on maximizing music's therapeutic benefits. The playlists will be purely instrumental, with a 60-80 bpm tempo, and feature melodies and harmonies designed for stress relief, including soothing, grounding, meditation, emotional release, etc. This approach is resource-efficient and easily accessible, allowing participants to integrate it into daily pain self-management strategies. Participants will be asked to engage in the MBI in the morning and at night for 30 minutes each, wearing the abdominal belt and smartwatch.
  Interventions: Behavioral: Music intervention

INTERVENTIONS:
Behavioral: Music intervention — Based on the NIH toolkit and MBIs reporting guidelines, the engagement in this pilot study will be receptive by providing participants with prerecorded, preselected playlists. Participants will also receive a guided video on maximizing music's therapeutic benefits. The playlists will be purely instrumental, with a 60-80 bpm tempo, and feature melodies and harmonies designed for stress relief, including soothing, grounding, meditation, emotional release, etc. This approach is resource-efficient and easily accessible, allowing participants to integrate it into daily pain self-management strategies. Participants will be asked to engage in the MBI in the morning and at night for 30 minutes each, wearing the abdominal belt and smartwatch.

SUMMARY:
The proposed pilot study aims to assess the underlying mechanisms of the MBI on IBS pain and the feasibility of using novel technology in the outcome measurements. The specific aims of this pilot mechanistic clinical trial are to:

1. . identify the mechanisms underlying the impact of MBI on IBS-related pain, stress responses, quantitative pain sensitivity, and gut microbiome profiles.
2. . evaluate the technological feasibility of using a wearable abdominal sensor belt and smartwatch system in measuring MBI impacts on pain in home settings.

Researchers will conduct a one-arm pre- and post-music intervention among patients with Irritable Bowel Syndrome, collect the IBS pain mechanistic biobehavioral markers, and analyze the underlying pathways of the music analgesic effect.

Participants will be asked to:

1. . engage in a 4-week intervention of 20 minutes, both during the day and at night, for at least five days per week.
2. . have two one-hour lab visits

DETAILED DESCRIPTION:
Purpose The proposed pilot study aims to assess the underlying mechanisms of the MBI on IBS pain and the feasibility of using novel technology in the outcome measurements. Irritable bowel syndrome (IBS) is the most common disorder of brain-gut interactions, characterized primarily by recurrent chronic abdominal pain, which severely impacts the quality of life and productivity of affected individuals, particularly women and young adults. Music-based interventions (MBIs) have shown promise in reducing pain cognitive processing and stress, potentially influencing pain perception in the brain and physiological arousal in the autonomic nervous system (ANS). Therefore, MBIs hold promising therapeutic potential for IBS pain management by targeting the overlapping mechanical pathways in the brain-gut axis (BGA).

Objectives The objective 1 is to identify the mechanisms underlying the impact of MBI on IBS-related pain, stress responses, quantitative pain sensitivity, and gut microbiome profiles.

The objective 2 is to evaluate the technological feasibility of using a wearable abdominal sensor belt and smartwatch system in measuring MBI impacts on pain in home settings.

Study Population In this pilot study, 30 participants with diagnosis of IBS will be recruited. The study focuses on this population because recurrent abdominal pain, discomfort, and altered bowel habits are the core clinical symptoms of patients with IBS. The prevalence of IBS is around 20% in the United States, with annual direct costs of care and indirect lost study/work productivity estimated at more than $21 billion in the United States.

Number of Participants Investigators plan to recruit 30 participants diagnosed with IBS for this pilot study. The sample size is based on investigators' prior experience and the recommended sample size for a pilot study to provide precise estimates.

Study Design This pilot mechanistic study is a one-arm pre- and post- intervention design. The pathways underlying neural and physiologic response to music and brain-gut interaction among IBS patients provide a cue to understand the complex interplay of outcome variables. Participants will be engaged in MBI for 20 minutes during the day and at night, at least five days a week, with the abdominal belt and smartwatch data acquisition during a four-week home-based intervention period. Throughout the study period, investigators will collect IBS pain mechanistic biobehavioral makers, including all real-time visceral pain indicators collected via the abdominal belt, real-time visual analog scale (VAS) pain report by smartwatch, and self-reported pain and stress status. Additionally, investigators will collect stool samples to investigate gut microbiome profiles and assess pain sensitivity through quantitative sensory testing (QST) equipment at two lab visits. Functional regression models and pathway analysis will determine the association between these factors.

Study Duration The pilot study will last for one year. Participants will attend two lab visits, each lasting approximately one hour. After the first lab visit, participants will be asked to engage in a music-based intervention using an abdominal belt and a smartwatch for 20 minutes, both during the day and at night, for at least five days per week. Weekly 15-minute meetings of the research assistants with each participant will be scheduled to follow up on issues encountered.

Outcome Variables Investigators will collect mechanistic biobehavioral markers of IBS pain, including real-time visceral pain indicators (electrodermal activity (EDA), electrocardiogram (ECG), and electromyogram (EMG)) via the abdominal belt, real-time visual analog scale (VAS) pain reports via the smartwatch, self-reported pain, stool samples, and quantitative pain sensitivity testing data. Additionally, investigators will assess participants' adherence to study protocols, completeness of data collection, and post-intervention satisfaction.

Locations/Facilities Participants' lab visits will take place at the Yale School of Nursing (YSN) Center for Biobehavioral Health Research and the Biobehavioral Research Laboratory (BBL). Research assistants will schedule weekly online meetings via Zoom with participants to gather feedback and address any issues encountered. Recruitment will be conducted through advertisements at collaborating gastrointestinal (GI) specialist offices and clinics affiliated with Yale New Haven Hospital. An advertising poster will be attached to bulletin boards on Yale west and main campus in order to draw attention from prospective participants.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 50 years old,
* can speak and read English,
* having a confirmed diagnosis of IBS from a healthcare provider,
* having experienced moderate pain (≥3 out of 10 on a numeric rating scale) at least four days a week for the past three months,
* be willing to participate in a 4-week intervention and attend two lab visits, and
* having daily access to an internet-enabled device for MBI.

Exclusion Criteria:

* having a severe psychiatric disorder requiring inpatient treatment in the past six months,
* regularly using opioids or illicit substances, or have used probiotics or antibiotics within two weeks prior to enrollment,
* having celiac disease, inflammatory bowel disease, or a history of major gastrointestinal surgery,
* concurrently participate in another IBS-related intervention study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
IBS visceral pain index | From intervention enrollment to the end of treatment at 4 weeks
  The sensitive objective integrated multimodal electrophysiological (OIME) index will be used as a biomarker for visceral pain evaluation, which will anticipate achieving robust and objective prediction of the pain level. Via machine learning and deep learning analysis, we will quantify the pain level based on key indices from time- and frequency-domain analysis of the objective EDA, ECG, and EMG recordings collected from the abdominal belt.
Real-time self-reported pain | From intervention enrollment to the end of treatment at 4 weeks
  The visual analog scale ranging from 0 (no pain) to 100 (highest level of pain) will be used to reflect the real-time episodes of visceral pain.
Brief Pain Inventory | through study completion, an average of 1 year
  The 9-item Brief Pain Inventory (BPI) scale sensitively assesses the severity of pain, the most painful area, the impact of pain on daily functions, medications, and the change in pain relief in the past 24 hours and the past week on a 0-10 (0= no pain or interference, 10= the worst possible pain or complete interference); A higher mean score indicates greater severity or interference. Cronbach alpha ranges from 0.77-0.91.
Pain sensitivity | through study completion, an average of 1 year
  We will assess participants' peripheral and central pain sensitivity using the comprehensive QST equipment established by the German Research Network on Neuropathic Pain as a protocol to examine thermal and mechanical sensory function44. The QST assessment includes (1) cutaneous mechanical pain sensitivity, which measures tolerance, threshold, temporal summation, and after-sensations; (2) heat and cold pain sensitivity, assessing threshold, tolerance, and ratings of supra-threshold stimuli; and (3) pressure pain thresholds. Quantifying sensory alterations in the IBS patient population offers insight into pain modulatory systems, both pain facilitation (hyperalgesia) and pain inhibition (hypoalgesia)
IBS-quality of life (IBS-QOL) | through study completion, an average of 1 year
  The IBS-QOL is a 34-item self-report questionnaire with a five-point Likert scale. It is specifically designed to measure the QOL in individuals with IBS. Total scores are calculated by adding up all the item responses, with higher scores indicating a better QOL. Psychometric evaluations have shown that the IBS-QOL is reliable, with a Cronbach's alpha of 0.96. It also demonstrates strong construct validity and is highly sensitive to detecting changes undergoing interventions.
16S rRNA Gene-based Analysis of Gut Microbiota | through study completion, an average of 1 year
  Our team has established the protocols for stool sample collection and processing and tested them in preliminary studies. Stool samples will be collected by a researcher-provided OMNIgene●GUT microbiome collection kit (DNA Genotek, Inc.); this easy self-collection system allows for stabilizing samples at room temperature for 14 days. RAs will provide adequate information and training to the participants about stool collection using the kits at in-person lab visits. Participants can return the samples to the repository by mail using a researcher-provided envelope. Samples will be immediately frozen upon collection at -80° C in the YSN BBL. Samples will be assigned a unique ID number, systematically entered into the specimen repository and database, and profiled by 16S rRNA Illumina sequencing. Paired-end 16S rRNA gene sequencing and analysis will be performed at the University of Connecticut Microbial Analysis, Resources, and Services (MARS) facility on an Illumina MiSeq system.

SECONDARY OUTCOMES:
Perceived Stress Scale-10 (PSS-10) | through study completion, an average of 1 year
  PSS-10 will be used to self-report the level of perceived stress in various life situations. It includes ten items rated on a 5-point scale, from "never" to "very often." The total score can range from 0 to 40, with a higher score indicating a higher stress level. The PSS has demonstrated high internal consistency and test-retest reliability.
Feasibility of using new technology in outcome measurements | From enrollment to the end of treatment at 4 weeks
  The feasibility of utilizing wearable devices for pain and stress measurement will be evaluated based on participant adherence to study protocols, data collection completeness, and participants' satisfaction. These data will provide insight into the practicality of integrating bio-signal monitoring technology in objective outcome measurements.
Intervention Adherence | through study completion, an average of 1 year
  Adherence will be tracked through the number of participants following the protocol over time, including daily usage patterns. Participants will log the frequency, timing, and duration of device usage in a structured online diary using the REDCap system.
Data recording completeness | through study completion, an average of 1 year
  Data recording completeness will be assessed by analyzing device synchronization and the proportion of missing data. Retention rates will be calculated based on participant continuity throughout the study duration.
Participant satisfaction | From intervention enrollment to the end of treatment at 4 weeks
  Post-intervention surveys will be administered to assess participant satisfaction, complemented by weekly feedback meetings to capture ongoing impressions and address any barriers to compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Weizi Wu, PhD, Principal Investigator — Yale School of Nursing; Xiaomei Cong, PhD, Principal Investigator — Yale School of Nursing
Locations (1):
- Yale School of Nursing, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
To ensure participant privacy and confidentiality, investigators will not share any individual participant data (IPD) with others. But this study is applying for an NIH U24 Pilot grant, which may have specific sharing requirements from the funding sponsor.

REFERENCES:
- [Result] Huang KY, Wang FY, Lv M, Ma XX, Tang XD, Lv L. Irritable bowel syndrome: Epidemiology, overlap disorders, pathophysiology and treatment. World J Gastroenterol. 2023 Jul 14;29(26):4120-4135. doi: 10.3748/wjg.v29.i26.4120. PMID 37475846
- [Result] Burns DS, Meadows AN, Althouse S, Perkins SM, Cripe LD. Differences between Supportive Music and Imagery and Music Listening during Outpatient Chemotherapy and Potential Moderators of Treatment Effects. J Music Ther. 2018 Mar 9;55(1):83-108. doi: 10.1093/jmt/thy001. PMID 29471518
- [Result] Burns DS, Perkins SM, Tong Y, Hilliard RE, Cripe LD. Music Therapy is Associated With Family Perception of More Spiritual Support and Decreased Breathing Problems in Cancer Patients Receiving Hospice Care. J Pain Symptom Manage. 2015 Aug;50(2):225-31. doi: 10.1016/j.jpainsymman.2015.02.022. Epub 2015 Apr 1. PMID 25839735
- [Result] Burns DS. Theoretical rationale for music selection in oncology intervention research: an integrative review. J Music Ther. 2012 Spring;49(1):7-22. doi: 10.1093/jmt/49.1.7. PMID 22803255
- [Result] Orock A, Yuan T, Greenwood-Van Meerveld B. Importance of Non-pharmacological Approaches for Treating Irritable Bowel Syndrome: Mechanisms and Clinical Relevance. Front Pain Res (Lausanne). 2021 Jan 21;1:609292. doi: 10.3389/fpain.2020.609292. eCollection 2020. PMID 35295688
- [Result] Black CJ, Ford AC. Best management of irritable bowel syndrome. Frontline Gastroenterol. 2020 May 28;12(4):303-315. doi: 10.1136/flgastro-2019-101298. eCollection 2021. PMID 34249316
- [Result] Cong X, Perry M, Bernier KM, Young EE, Starkweather A. Effects of Self-Management Interventions in Patients With Irritable Bowel Syndrome: Systematic Review. West J Nurs Res. 2018 Nov;40(11):1698-1720. doi: 10.1177/0193945917727705. Epub 2017 Aug 30. PMID 28854852
- [Result] Lembo A, Sultan S, Chang L, Heidelbaugh JJ, Smalley W, Verne GN. AGA Clinical Practice Guideline on the Pharmacological Management of Irritable Bowel Syndrome With Diarrhea. Gastroenterology. 2022 Jul;163(1):137-151. doi: 10.1053/j.gastro.2022.04.017. PMID 35738725
- [Result] Arnold CA, Bagg MK, Harvey AR. The psychophysiology of music-based interventions and the experience of pain. Front Psychol. 2024 May 10;15:1361857. doi: 10.3389/fpsyg.2024.1361857. eCollection 2024. PMID 38800683
- [Result] de Witte M, Spruit A, van Hooren S, Moonen X, Stams GJ. Effects of music interventions on stress-related outcomes: a systematic review and two meta-analyses. Health Psychol Rev. 2020 Jun;14(2):294-324. doi: 10.1080/17437199.2019.1627897. Epub 2019 Jul 15. PMID 31167611
- [Result] Chen WG, Iversen JR, Kao MH, Loui P, Patel AD, Zatorre RJ, Edwards E. Music and Brain Circuitry: Strategies for Strengthening Evidence-Based Research for Music-Based Interventions. J Neurosci. 2022 Nov 9;42(45):8498-8507. doi: 10.1523/JNEUROSCI.1135-22.2022. PMID 36351825
- [Result] Mayer EA, Ryu HJ, Bhatt RR. The neurobiology of irritable bowel syndrome. Mol Psychiatry. 2023 Apr;28(4):1451-1465. doi: 10.1038/s41380-023-01972-w. Epub 2023 Feb 2. PMID 36732586